CLINICAL TRIAL: NCT00780793
Title: Effect of TNF-blocker Injections Spacing on Rheumatoid Arthritis Inflammatory Activity in Patients in Clinical Remission or Low Disease Activity
Brief Title: Spacing of TNF-blocker Injections in Rheumatoid Arthritis Study
Acronym: STRASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Society of Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOM 07127
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2008-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Remission; Therapeutic strategy; DMARDs; Biological agents
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-M : Maintenance (Active Comparator): Usual care
  Interventions: Drug: DMARD maintenance
- 2 -S : Spacing of TNF-blocker injections (Experimental): Spacing of TNF-blocker injections
  Interventions: Drug: progressive spacing of TNF-blocker injections

INTERVENTIONS:
Drug: progressive spacing of TNF-blocker injections — Experimental arm
  Progressive spacing of TNF-blocker injections according to the following algorithm :
  * if DAS28 ≤ 2.6 at trimestrial assessment: go for step N+1
  * if DAS28 > 2.6 and DAS28 change ≤ 0.6: continue at step N
  * if DAS28 > 2.6 and DAS28 change > 0.6 : return to step N-1 (relapse as defined by the European expert consensus).
  Step 0 (inclusion) :
  * Adalimumab 40 mg / 14 days
  * Etanercept 50 mg / 7 days
  Step 1 :
  * Adalimumab 40 mg / 21 days
  * Etanercept 50 mg / 10 days
  Step 2 :
  * Adalimumab 40 mg / 28 days
  * Etanercept 50 mg / 14 days
  Step 3 :
  * Adalimumab 40 mg / 42 days
  * Etanercept 50 mg / 21 days
  Step 4 :
  * TNF-blocker stop
  Other Names: Spacing (S)
  Arms: 2 -S : Spacing of TNF-blocker injections
Drug: DMARD maintenance — DMARD maintenance
  Arms: 1-M : Maintenance

SUMMARY:
Remission is nowadays the recommended therapeutic objective in rheumatoid arthritis. Once this objective is achieved thanks to TNF-blockers, the optimal therapeutic strategy remains unclear, either therapeutic maintenance or progressive DMARD tapering (with a non quantified risk of disease flare).

STRASS is a 2-arm randomized controlled trial aiming to compare these 2 strategies (DMARD maintenance or progressive spacing of TNF-blocker injections) in terms of remission maintenance, relapse risk, safety issues and economic consequences during 18 months.

The inclusion period is 18 months, between September 2008 and February 2010.

DETAILED DESCRIPTION:
Rationale:

Clinical remission is the therapeutic objective in rheumatoid arthritis, as recommended by professional practice guidelines. Once this objective is achieved with subcutaneous TNF-blockers, the maintenance of such treatments - highly efficacious but expensive and potentially toxic - is debated. To date, no reliable data are available to estimate the risk - benefice ratio associated with either their maintenance or their tapering.

Objectives:

In RA patients in remission, the study aims:

1. To compare RA inflammatory activity based on repeated measures of the Disease Activity Score (DAS) depending on 2 therapeutic schemes: (M) maintenance of unchanged TNF-blockers or (S) tapering of TNF-blocker doses by progressive spacing of subcutaneous injections according to a predefined algorithm;
2. To estimate the cost - effectiveness ratio of TNF-blocker spacing as compared to TNF-blocker maintenance.

Inclusion criteria:

* Patients aged 18 or more, diagnosed with RA according to the 1987 ACR classification criteria;
* RA treated with subcutaneous TNF-blockers (etanercept or adalimumab) at stable and standard dosage for 1 year or more, as monotherapy or associated with stable conventional DMARD;
* RA in clinical remission, defined as a stable DAS28 ≤ 2.6 for 6 months or more, without any structural damage progression on X-rays (local reading by the treating rheumatologist);

Exclusion criteria:

* Treatment with steroids;
* progressing disease on X-rays during the year preceding the trial;
* surgery planed in the 18 coming months;
* pregnancy;
* on-going neoplastic disease;
* other auto-immune disorders different from RA;
* inability to speak or understand French;
* absence of signed informed consent;
* absence of medical insurance coverage.

Sample size calculation: 250 patients, 125 for each arm.

Centers: 22 inclusion centers in France.

Research duration: 3 years. Participation duration for each patient: 18 months. Inclusion period duration: 18 months (Sep 2008 - Feb 2010).

Methods:

Equivalence trial, prospective, randomized, controlled versus usual care, patients remaining blinded of the tested hypotheses.

Investigators assessing disease activity remain blind of the protocol arm. The statistical analysis will be based on a mixed linear model taking into account repeated data.

Randomization:

Computer-assisted randomization (CleanWeb software) by blocks of unequal size, stratified on inclusion centers and TNF-blocker molecule.

Primary endpoint:

RA inflammatory activity over 18 months estimated by DAS28 repeated measures.

Secondary endpoints:

* RA inflammatory activity over 18 months estimated by DAS44 repeated measures;
* Cost - Effectiveness ratio calculated as: (CostMaintenance - CostSpacing) / (EfficacyMaintenance - EfficacySpacing);
* Relapse rate over 18 months based on Kaplan Meier survival analysis;
* Functional impairment based on HAQ index;
* Health-related quality of life on SF-36;
* Utility based on EQ-5D instrument;
* Structural damage progression over 18 months assessed with the van der HEIJDE-modified Sharp score (SHS);
* Safety;
* Determinants of maintained remission or relapse after TNF-blocker injection spacing.

Research time sheet:

Clinical, biological and imaging follow-up is based on guidelines-recommended RA follow-up.

Biological work-ups specifically dedicated to the research represent 80 mL. The others are part of usual care and may be performed in non-hospital laboratories.

Expected results and perspectives:

The trial aims to test the feasibility and the risk - benefit ratio of a step-down strategy for TNF-blockers in the course of RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more, diagnosed with RA according to the 1987 ACR classification criteria;
* RA treated with subcutaneous TNF-blockers (étanercept or adalimumab) at stable and standard dosage for 1 year or more, as monotherapy or associated with stable conventional DMARD;
* RA in clinical remission, defined as a stable DAS28 ≤ 2.6 for 6 months or more, without any structural damage progression on X-rays (local reading by the treating rheumatologist);

Exclusion Criteria:

* Treatment with steroids;
* progressing disease on X-rays during the year preceding the trial;
* surgery planed in the 18 coming months;
* pregnancy;
* on-going neoplastic disease;
* other auto-immune disorders different from RA;
* inability to speak or understand French;
* absence of signed informed consent;
* absence of medical insurance coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
RA inflammatory activity over 18 months based on repeated DAS28 measures | over 18 months

SECONDARY OUTCOMES:
RA inflammatory activity over 18 months estimated by DAS44 repeated measures | over 18 months
Cost - Effectiveness ratio calculated as: (CostMaintenance - CostSpacing) / (EfficacyMaintenance - EfficacySpacing); | during the study
Relapse rate over 18 months based on Kaplan Meier survival analysis | over 18 months
Functional impairment based on HAQ index | during the study
Health-related quality of life on SF-36 | during the study
Utility based on EQ-5D instrument | during the study
Structural damage progression over 18 months assessed with the van der HEIJDE-modified Sharp score (SHS) | over 18 months
Determinants of maintained remission or relapse after TNF-blocker injection spacing | during teh study

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fautrel, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de rhumatologie / Groupe hospitalier Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Fautrel B, Pham T, Alfaiate T, Gandjbakhch F, Foltz V, Morel J, Dernis E, Gaudin P, Brocq O, Solau-Gervais E, Berthelot JM, Balblanc JC, Mariette X, Tubach F. Step-down strategy of spacing TNF-blocker injections for established rheumatoid arthritis in remission: results of the multicentre non-inferiority randomised open-label controlled trial (STRASS: Spacing of TNF-blocker injections in Rheumatoid ArthritiS Study). Ann Rheum Dis. 2016 Jan;75(1):59-67. doi: 10.1136/annrheumdis-2014-206696. Epub 2015 Jun 23. PMID 26103979